CLINICAL TRIAL: NCT06618378
Title: Effectiveness of Biofeedback Training in Children with Neurogenic Bladder and Bowel Disorder with Spina Bifida
Brief Title: Effectiveness of Biofeedback Training in Children with Neurogenic Bladder and Bowel Disorder Wıth Spina Bifida
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Fatma Nur Erçetin, Physiotherapist, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neurogenic Bladder
Record Dates: First submitted 2024-06-05; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Spina Bifida
Keywords: spina bifida; biofeedback; urotherapy; neurogenicbladder
MeSH Terms: conditions — Spinal Dysraphism | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: There will be 3 groups followed at the same time.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention)
- Urotherapy educational group (Active Comparator)
  Interventions: Behavioral: urotherapy educational group
- Biofeedback exercise group combined with breathing exercise (Experimental)
  Interventions: Behavioral: Biofeedback exercise combined with breathing exercise; Behavioral: urotherapy educational group

INTERVENTIONS:
Behavioral: Biofeedback exercise combined with breathing exercise — Urotherapy training will be given at the beginning of the treatment process. Contraction and relaxation will be applied around the external sphincter in combination with diaphragmatic breathing by visual imagery with EMG biofeedback application. The second channel EMG will be placed on the transversus abdominus muscle and its activation will be checked. The treatment will be completed with 30-minute sessions twice a week for 12 weeks. Each session will consist of 40 cycles of 10 minutes of diaphragmatic breathing exercise followed by 20 minutes of 10 seconds of contraction followed by 20 seconds of relaxation.
  Arms: Biofeedback exercise group combined with breathing exercise
Behavioral: urotherapy educational group — 1. An important part of urotherapy is to provide parents and children with detailed explanations of etiology, prevalence and pathophysiology. This will reassure parents and help them understand the causes of the child's bedwetting accidents and the rationale for treatment. This will increase compliance with treatment.
  2. Recommendations are given regarding appropriate fluid intake and regular voiding throughout the day. The child is encouraged to go to the toilet seven times a day and drink seven glasses of water.
  3. The correct sitting position for the toilet is explained. If the feet do not touch the floor easily, it is recommended to use a step stool for foot support. Additionally, children are taught to relax their abdomen when peeing.
  4. In addition to monitoring and motivation, a bladder diary should be kept to give the child and parents an idea about the progress of treatment, compliance with treatment and continuity.
  Arms: Biofeedback exercise group combined with breathing exercise; Urotherapy educational group

SUMMARY:
The aim of this study is to examine and compare the bladder and bowel functions, activation of pelvic floor and abdominal muscle groups and quality of life of children diagnosed with spina bifida who did not receive any treatment due to bladder-intestinal dysfunction, received only urotherapy training and received biofeedback training combined with breathing.

The type of study is clinical trial. Question 1: Does biofeedback training combined with breathing have an effect on bladder and bowel functions, activation of pelvic floor and abdominal muscle groups and quality of life in spina bifida patients with neurogenic bladder and bowel disorders? Question 2: Does urotherapy training have an effect on bladder and bowel functions, activation of pelvic floor and abdominal muscle groups and quality of life in spina bifida patients with neurogenic bladder and bowel disorders? Group 1: control group Group 2: urotherapy training group Group 3: Biofeedback exercise training group combined with breathing There will be no extra treatment to group 1. Urotherapy Training: Standard urotherapy is a combined method that includes clinical assessment (recording voiding frequencies, voiding volumes and incontinence episodes in a bladder diary), voiding habit training, behavior modification instructions, lifestyle recommendations regarding fluid intake and supporting children and their parents through the process.

Exercise Training: Urotherapy training will be given at the beginning of the treatment process. Contraction and relaxation will be applied around the external sphincter in combination with diaphragmatic breathing by visual imagery with EMG biofeedback application.

Group 1, group 2 and group 3 will be compared.

DETAILED DESCRIPTION:
To the best of our knowledge, no study has been found in which biofeedback training combined with breathing was applied on children with neurogenic bladder. Additionally, to the best of our knowledge, no study has been found in which biofeedback exercises were applied to children with spina bifida. Therefore, in this study, researchers aim to compare the bladder functions, pelvic floor and abdominal muscle activations and quality of life of children with spina bifida who do not have access to any alternative treatment, receive only urotherapy training and biofeedback training combined with breathing.The aim of this study is to examine and compare the bladder and bowel functions, activation of pelvic floor and abdominal muscle groups, and quality of life of children diagnosed with spina bifida who did not receive any treatment due to bladder-intestinal dysfunction, received only urotherapy training, and received biofeedback training combined with breathing.

Evaluation Methods Gross Motor Function Classification System (GMFCS): The basic scale used to classify mobility is the classification called Gross Motor Function Classification System (GMFCS). According to this classification, patients are divided into 5 groups, from level 1, who can walk without any problems, to level 5, who is wheelchair-bound.

General Headings of Each Level:

Level i: walks without restriction. Level ii: walks with restrictions. Level iii: walks using hand-held mobility devices. Level iv: self-motion is limited. Can use motorized mobility device. Level v: transported in a manually propelled wheelchair. Bladder and bowel diary: It is a form recorded by the child or his/her parents in a 48-hour period, in which the child daily schedule records the amount of fluid he/she takes in and excretes, the frequency of urination, the frequency of urinary incontinence, the activity in which the incontinence occurs, the stool he/she makes throughout the day, and the quality of the stool.

Voiding Disorders Symptom Score (VBSS): Voiding Disturbances Symptom Score (VBSS), which was developed by Akbal et al. and whose validity and reliability have been proven, includes 14 questions. The first 13 questions examine the child urinary and defecation habits, daytime and/or nighttime urinary incontinence, and urination functions; The 14th question is intended to evaluate the child general quality of life. In the evaluation of IBSS 1,2 and the 3rd question will receive a minimum of 0 and a maximum of 9 points; Min 0, max 5 points from the 4th question; Min 0, max 2 points from Questions 5, 8, 9, 11, 12 and 13; A minimum of 0 and a maximum of 33 points can be obtained from the scale, with a minimum of 0 and a maximum of 3 points from the 6th Question and a minimum of 0 and a maximum of 1 from the 7th and 10th Questions. Although the Cronbach Alpha value of the scale is 0.50, the Cronbach Alpha value for this study was determined as 0.711.

Superficial EMG: According to the International Continence Society (ICS), electromyography (EMG) should be performed before LUTD treatment. Pelvic floor and abdominal muscle activation was performed with the same device (NeuroTrac myoplus 4, Verity Medical Ltd, UK), which can take measurements from two different channels at the same time. Activation will be checked at the initial and final evaluation and before each biofeedback exercise training to determine the condition of the pelvic floor and abdominal muscles. With EMG, muscle strength, endurance, speed, coordination, oscillation and relaxation time data will be recorded.

Quality of life measure for children (PedQL): The Pediatric Quality of Life Inventory (Children Hospital and Health Center, San Diego, California) is a modular instrument used to measure health-related quality of life (HRQOL) in children and adolescents ages 2 to 18 years. PedsQL 4.0 Generic Core Scales are multidimensional child self-report and parent proxy report scales developed as generic core measures to be integrated with PedsQL Disease-Specific Modules. The PedsQL 4.0 Generic Core Scales consist of 23 items valid for healthy school and community populations as well as pediatric populations with acute and chronic health conditions.

Educational Programs Urotherapy Training: Standard urotherapy is a combined method that includes clinical assessment (recording voiding frequencies, voiding volumes, and incontinence episodes in a bladder diary), voiding habit training, behavior modification instructions, lifestyle recommendations regarding fluid intake, and supporting children and their parents through the process.

1. An important part of urotherapy is to provide parents and children with detailed explanations of etiology, prevalence and pathophysiology. This will reassure parents and help them understand the causes of the child's bedwetting accidents and the rationale for treatment. This will increase compliance with treatment.
2. Recommendations are given regarding appropriate fluid intake and regular voiding throughout the day. The child is encouraged to go to the toilet seven times a day and drink seven glasses of water.
3. The correct sitting position for the toilet is explained. If the feet do not touch the floor easily, it is recommended to use a step stool for foot support. Additionally, children are taught to relax their abdomen when peeing.
4. In addition to monitoring and motivation, a bladder diary should be kept to give the child and parents an idea about the progress of treatment, compliance with treatment and continuity.

Exercise Training: Urotherapy training will be given at the beginning of the treatment process. Contraction and relaxation will be applied around the external sphincter in combination with diaphragmatic breathing by visual imagery with EMG biofeedback application. The second channel EMG will be placed on the transversus abdominus muscle and its activation will be checked. The treatment will be completed with 30-minute sessions twice a week for 12 weeks. Each session will consist of 40 cycles of 10 minutes of diaphragmatic breathing exercise followed by 20 minutes of 10 seconds of contraction followed by 20 seconds of relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with meningomyelocele type spina bifida
* Individuals between the ages of 5-18.

Exclusion Criteria:

* Presence of lower urinary tract infection
* Presence of abdominal surgery in the last 3 months.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-21 (Estimated); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
The effect of biofeedback training combined with breathing on bladder and bowel functions in spina bifida patients with neurogenic bladder and bowel disorders. | 3 months
  The primary outcome measure will be assessed by Voiding Disorders Symptom Score . The lowest score is 34, while the highest score is 170. Scale Evaluation: An increase in the total score obtained from the scale indicates an increase in the quality of life of individuals related to the disease.
The effect of biofeedback training combined with breathing on quality of life in spina bifida patients with neurogenic bladder and bowel disorders. | 3 months
  The primary outcome measure will be assessed by The Pediatric Quality of Life Inventory (PedQL). In the inventory prepared according to the five-point Likert system, 0 = Never causes a problem, 1 = Almost never causes a problem, 2 = Sometimes causes a problem, 3 = Often causes a problem and 4 = Always causes a problem. A linear conversion is applied in the calculation of the total score of the scale and it turns into 0-100 points. As the score decreases, the quality of life increases.
The effect of biofeedback training combined with breathing on activation of abdominal muscle groups in spina bifida patients with neurogenic bladder and bowel disorders. | 3 months
  The primary outcome measure will be assessed by superficial electromyography (EMG) outcomes. With the EMG device, the maximal, average and minimum contraction stimulation frequencies of the muscles and the maximal voluntary contraction percentage data will be obtained. The measurements will be taken by placing the channel around the transversus abdominus muscle (two fingers above and medial to the anterior superior iliac spine).
The effect of biofeedback training combined with breathing on activation of pelvic floor muscle groups in spina bifida patients with neurogenic bladder and bowel disorders. | 3 months
  The primary outcome measure will be assessed by superficial electromyography (EMG) outcomes. With the EMG device, the maximal, average and minimum contraction stimulation frequencies of the muscles and the maximal voluntary contraction percentage data will be obtained. The measurements will be taken by placing the first channel around the external sphincter at 2-7 clock.

SECONDARY OUTCOMES:
The effect of urotherapy training on bladder and bowel functions in spina bifida patients with neurogenic bladder and bowel disorders. | 3 months
  The primary outcome measure will be assessed by Voiding Disorders Symptom Score . The lowest score is 34, while the highest score is 170. Scale Evaluation: An increase in the total score obtained from the scale indicates an increase in the quality of life of individuals related to the disease.
The effect of urotherapy training on quality of life in spina bifida patients with neurogenic bladder and bowel disorders. | 3 months
  The primary outcome measure will be assessed by The Pediatric Quality of Life Inventory (PedQL). In the inventory prepared according to the five-point Likert system, 0 = Never causes a problem, 1 = Almost never causes a problem, 2 = Sometimes causes a problem, 3 = Often causes a problem and 4 = Always causes a problem. A linear conversion is applied in the calculation of the total score of the scale and it turns into 0-100 points. As the score decreases, the quality of life increases.
The effect of urotherapy training combined with breathing on activation of abdominal muscle groups in spina bifida patients with neurogenic bladder and bowel disorders. | 3 months
  The primary outcome measure will be assessed by superficial electromyography (EMG) outcomes. With the EMG device, the maximal, average and minimum contraction stimulation frequencies of the muscles and the maximal voluntary contraction percentage data will be obtained. The measurements will be taken by placing the channel around the transversus abdominus muscle (two fingers above and medial to the anterior superior iliac spine).
The effect of urotherapy training on activation of pelvic floor muscle groups in spina bifida patients with neurogenic bladder and bowel disorders. | 3 months
  The primary outcome measure will be assessed by superficial electromyography (EMG) outcomes. With the EMG device, the maximal, average and minimum contraction stimulation frequencies of the muscles and the maximal voluntary contraction percentage data will be obtained. The measurements will be taken by placing the first channel around the external sphincter at 2-7 clock.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Nur Erçetin, MSc, Principal Investigator — Doctoral thesis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu L, Fu C, Zhang Q, Xiong F, Peng L, Liang Z, Chen L, He C, Wei Q. Efficacy of biofeedback, repetitive transcranial magnetic stimulation and pelvic floor muscle training for female neurogenic bladder dysfunction after spinal cord injury: a study protocol for a randomised controlled trial. BMJ Open. 2020 Aug 5;10(8):e034582. doi: 10.1136/bmjopen-2019-034582. PMID 32759239
- [Background] Zivkovic VD, Stankovic I, Dimitrijevic L, Kocic M, Colovic H, Vlajkovic M, Slavkovic A, Lazovic M. Are Interferential Electrical Stimulation and Diaphragmatic Breathing Exercises Beneficial in Children With Bladder and Bowel Dysfunction? Urology. 2017 Apr;102:207-212. doi: 10.1016/j.urology.2016.12.038. Epub 2016 Dec 28. PMID 28040503
- [Background] Libo LM, Arnold GE, Woodside JR, Borden TA, Hardy TL. EMG biofeedback for functional bladder-sphincter dyssynergia: a case study. Biofeedback Self Regul. 1983 Jun;8(2):243-53. doi: 10.1007/BF00998854. PMID 6357288